CLINICAL TRIAL: NCT01956786
Title: Efficacy of Amlodipine-Folic Acid Tablets on Reduction of Blood Pressure and Plasma Homocysteine in Patients With Mild to Moderate Hypertension, Hyperhomocysteinemia and Angiotension-Converting Enzyme Inhibitor Intolerance
Brief Title: Efficacy of Amlodipine-Folic Acid Tablets on Reduction of Blood Pressure and Plasma Homocysteine
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Ausa Pharmed Co.,Ltd (Industry)
Collaborators: Ruijin Hospital (Other); Second Affiliated Hospital of Nanchang University (Other); Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ausa-Amlodipine B
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-07

CONDITIONS: Essential Hypertension
Keywords: Amlodipine; Folic Acid; Homocysteine; Blood Pressure
MeSH Terms: conditions — Essential Hypertension | interventions — Contraceptives, Oral; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Amlodipine (Active Comparator): 5mg amlodipine,once daily for 8 weeks
  Interventions: Drug: Amlodipine
- Amlodipine-FA tablet,low dose group (Experimental): 5mg amlodipine combined with 0.4mg of folic acid (FA),once daily for 8 weeks.
  Interventions: Drug: Amlodipine-FA tablet,low dose group
- Amlodipine-FA tablet,high dose group (Experimental): 5mg amlodipine combined with 0.8mg of folic acid (FA),once daily for 8 weeks.
  Interventions: Drug: Amlodipine-FA tablet,high dose group

INTERVENTIONS:
Drug: Amlodipine-FA tablet,low dose group — 5mg amlodipine combined with 0.4mg folic acid,once daily (Low-dose group)
  Other Names: low dose
  Arms: Amlodipine-FA tablet,low dose group
Drug: Amlodipine-FA tablet,high dose group — 5mg amlodipine combined with 0.8mg folic acid,once daily (High-dose group)
  Other Names: high dose
  Arms: Amlodipine-FA tablet,high dose group
Drug: Amlodipine — 5mg amlodipine,once daily
  Other Names: control
  Arms: Amlodipine

SUMMARY:
To evaluate the efficacy of Amlodipine-Folic Acid Tablets on reduction of blood pressure and plasma total homocysteine.

DETAILED DESCRIPTION:
Traditional risk factors are estimated to account for only part of cardiovascular disease (CVD)risk. Non-traditional risk factors such as increased homocysteine concentrations are believed to be causally related to CVD. The interactive effect between hypertension and hyperhomocysteinemia on the risk of CVD has received great attention. Methylenetetrahydrofolate reductase (MTHFR)was the main regulatory enzymes for homocysteine metabolism. MTHFR converts 5,10-methylene-THF into 5-methyl-THF. Polymorphism of MTHFR C677T leads to a reduction in enzyme activity, which may lead to an increased concentration of plasma homocysteine and lower levels of serum folate, particularly in those with low folate intake. Enalapril Maleate-Folate Tablets, known to reduce both blood pressure and serum homocysteine and thereby preventing stroke, was found to have adverse events, such as cough, called ACEI-intolerance in some patients.

In the present study, we sought to assess:(1)the efficacy and safety of Amlodipine-Folic Acid Tablets in lowing blood pressure and homocysteine in patients with mild to moderate hypertension, hyperhomocysteinemia (hcy≥10μmol/L)and ACEI intolerance;(2)whether the blood pressure and homocysteine-lowing efficacy of Amlodipine-Folic Acid Tablets can be modified by individual MTHFR C677T polymorphisms.

In all, about 540 patients with mild to moderate hypertension, hyperhomocysteinemia and ACEI intolerance will be enrolled in this trial. Eligible subjects are randomly and double-blindly assigned to one of the three treatment groups:1)amlodipine tablet(5mg,control group);2)amlodipine-folic acid tablet(5mg amlodipine combined with 0.4mg of folic acid,low FA group);or 3)amlodipine-folic acid tablet (5mg amlodipine combined with 0.8mg of folic acid,high FA group),once daily for 8 weeks.

The allocation of participants was programmed by an independent statistical coordinating center,encrypted,and sent to each study center.Tablet containers were labeled only with the name of the trial and the allocated concealment number.The participants,care partners,and all staff directly involved in the trial were blinded to interventions during the period of the trial.

Demographic and clinical information were obtained at baseline. Blood pressure was examined at baseline and every two weeks for a total period of 8 weeks. Blood homocysteine and folate concentrations were examined at baseline and at 4th、8th weeks of the trial. MTHFR C677T genotypes were determined for each study subject.

All analyses will be performed according to the principle of intention to treat.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years;
2. Sedentary systolic blood pressure between 140 mmHg and 180 mmHg, and/or sedentary diastolic blood pressure between 90 mmHg and 110 mmHg;
3. Plasma homocysteine ≥ 10μmol/L;
4. ACEI-intolerance
5. Signed the written informed consent.

Exclusion Criteria:

1. Pregnant women or women within lactation period;
2. Hypersensitive to Calcium Channel Blocker (CCB) or folic acid;
3. Easily hypersensitiveness;
4. Diagnosed secondary hypertension or skeptical secondary hypertension;
5. Severe hypertension (sedentary systolic blood pressure greater than or equal to 180 mmHg and/or sedentary diastolic blood pressure greater than or equal to 110 mmHg)
6. Severe diseases:

   1. Cardiovascular system:Diagnosed cardia insufficiency (New York Health Association [NYHA] Ⅲ level and higher);Hypertrophic obstructive cardiomyopathy (HOCM);Clinical significantly Valvular Disease of the Heart (VDH);Acute coronary syndrome or coronary artery interventional therapy or coronary artery bypass graft within three months;Severe arrhythmia such as atrial flutter, atrial fibrillation, atrioventricular block above Ⅱlevel, et al;
   2. Alimentary system:Active virus hepatitis;Any of alanine aminotransferase (ALT), aspartate aminotransferase (AST), galactosylhydroxylysyl glucosyltransferase (GGT), alkaline phosphatase (ALP), total bilirubin (TBIL), Direct Bilirubin (DB) was above 2 times of it's normal value upper limit, albumin (ALB) greater than 30 g/L;Stomach bulk resect and gastrojejunostomy;Stomach intestine malabsorption;
   3. Urinary system:Serum creatinine greater than or equal to 200 mmol/L;Diagnosed stenosis of renal artery, solitary kidney;Renal transplantation;
   4. Endocrine system:Type 1 diabetes mellitus or uncontrolled type 2 diabetes mellitus (fasting glucose greater than or equal to 11.1 mmol/L);Diagnosed and uncontrolled hyperthyrosis;
   5. Respiratory system:Pulmonary Heart Disease;Chronic Obstructive Pulmonary Disease(COPD);
   6. Neuropsychiatric system:Transient Ischemia Attach (TIA) or stroke within 3 months;Severe peripheral nerve or vegetative nerve functional disturbance; Psyche or nervous system dysfunction;Drugs or alcohol dependence;
   7. Others:Malignant tumor, malnutrition, haematogenesis dysfunction, et al;
7. Obviously abnormal laboratory examination or signs;
8. Taking other antihypertensive drugs and unwilling to stop;
9. Taking folic acid or other Vitamin B groups and unwilling to stop;
10. Ever to participant in any drug trial not yet approved within 4 weeks before the first visit.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2013-09; Primary Completion 2013-12 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Combined effective rate of blood pressure and plasma homocysteine reduction | Blood pressure was examined at baseline and every 2 weeks for a total period of 8 weeks.Blood homocysteine concentrations were measured at baseline and at 4th and 8th week of the trial.

SECONDARY OUTCOMES:
Blood pressure reduction or plasma homocysteine reduction | Blood pressure was examined at baseline and every 2 weeks of a total period of 8 weeks. Blood homocysteine concentrations was examined at baseline and at 4th and 8th week of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Jiguang, MD, Principal Investigator — Ruijin Hospital, Shanghai Jiao Tong University
Locations (3):
- China (3):
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Ruijin Hospital, Shanghai Jiao Tong Univesity, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Bao H, Huang X, Li P, Sheng C, Zhang J, Wang Z, Song D, Hu L, Ding C, Cheng Z, Yao C, Chen G, Cui Y, Qin X, Tang G, Wang X, Huo Y, Cheng X, Wang J. Combined use of amlodipine and folic acid are significantly more efficacious than amlodipine alone in lowering plasma homocysteine and blood pressure among hypertensive patients with hyperhomocysteinemia and intolerance to ACEI: A multicenter, randomized, double-blind, parallel-controlled clinical trial. J Clin Hypertens (Greenwich). 2023 Aug;25(8):689-699. doi: 10.1111/jch.14697. Epub 2023 Jul 11. PMID 37433173